CLINICAL TRIAL: NCT02970565
Title: Family Nurture Intervention, A Group Model: Short and Long Term Effects on Behavior and Development of Preschool Aged Children
Brief Title: Family Nurture Intervention, A Group Model in Connecticut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Martha G Welch, Associate Professor of Psychiatry (in Pediatrics and Pathology and Cell Biology), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AAAQ9547
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Behavior Problem; Development Delay; Emotional Disturbance; Family Conflict
Keywords: Family Nurture Intervention; Martha G. Welch MD; Randomized Control Trial; Pre-school Intervention; Preschool Intervention; Multiple Family Group Intervention; Emotional Connection; Co-regulation
MeSH Terms: conditions — Mental Disorders; Learning Disabilities; Affective Symptoms | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrition and Play Intervention (Experimental): Mother-child dyads who are enrolled into the study will be randomly assigned to the Nutrition and Play Intervention group.
  Interventions: Behavioral: Nutrition and Play Intervention
- Family Nurture Intervention (Experimental): Mother-child dyads who are enrolled into the study will be randomly assigned to the Family Nurture Intervention group.
  Interventions: Behavioral: Family Nurture Intervention

INTERVENTIONS:
Behavioral: Family Nurture Intervention — The mother-child pair will be asked to talk and play with each other as they customarily do. If the child becomes restless and dysregulated the mother will be coached by the Nurture Specialist to bring the child back into a calm state through sustained physical contact, comfort touch, soothing words, and eye contact.
  Other Names: FNI
  Arms: Family Nurture Intervention
Behavioral: Nutrition and Play Intervention — Mothers and children in the Play and Nutrition group will play educational and nutrition-focused games.
  Other Names: NPI
  Arms: Nutrition and Play Intervention

SUMMARY:
The purpose of this current study is to investigate the efficacy of a group model of Family Nurture Intervention in ameliorating behavioral problems in preschool-aged children. The behavioral, neurobiological and clinical insights gained from this project may eventually lead to better treatment of emotional, behavioral and developmental disorders. The investigator hypothesizes that the children who are treated with Family Nurture Intervention (FNI), which incorporates interactive touch with vocal soothing, and family practice in comforting, will show increased emotional connection and mother child co-regulation with better results in the outcome measures in the short term and long term.

DETAILED DESCRIPTION:
There are several early intervention programs that are available for children with emotional, behavioral and developmental disorders, ranging from behavioral treatment and sensory exposure therapy to pharmaceutical treatments. Although improvements in behavior have resulted from these interventions, they are limited in numerous ways. They are usually time-consuming, both for the child and the teacher or clinician providing the intervention. In order to see an effect of the intervention, most children must engage in the intervention procedure for several years. Moreover, the effects of most current intervention procedures are minimal to moderate. Pharmaceutical prescriptions are often accompanied by undesirable side effects that may modulate behavior, emotion, and physiological functions. The behavioral, neurobiological and clinical insights gained from this project may eventually lead to better treatment of emotional, behavioral and developmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Child is a singleton
* Mother can speak in English or Spanish
* Child is between the ages of 2 to 4 ½ years at date of enrollment
* Mother is 18 years of age or older at the time of consent
* Child demonstrates developmental deficit as measured by the SDQ (cutoff of 13 or more on the total score excluding the pro-social questions; OR 4 or less on the pro-social questions, which are reverse scored i.e. higher is better)
* Child must reside with mother

Exclusion Criteria:

* The child has severe congenital anomalies or chromosomal anomalies including Downs syndrome and Cerebral Palsy
* The child has a diagnosis of Autism
* The child has severe motor or physical disability
* Mother currently presents with psychosis or is currently taking antipsychotic medication
* Current maternal drug and/or alcohol abuse
* Mother has any current involvement with Child Protective Services (Department of Children and Families)
* Mother is pregnant
* Mother and/or infant has a medical condition or contagion that precludes intervention components

Ages: 24 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in Childhood Behavior Checklist (CBCL) Score | Baseline, 6 months
  The Childhood Behavior Checklist (CBCL) is a device by which parents or other individuals who know the child well rate a child's problem behaviors and competencies. This instrument can either be self-administered or administered through an interview. The CBCL can also be used to measure a child's change in behavior over time or following a treatment. The first section of this questionnaire consists of 20 competence items and the second section consists of 120 items on behavior or emotional problems.

SECONDARY OUTCOMES:
Co-regulation of Vagal Tone | Up to 12 months
  Using ECG data obtained during each follow-up visit, the investigators will characterize various parameters of cardiac function and regulation including assessments of parasympathetic modulation of heart rate. Long term individual differences in attention and emotional regulation are correlated with these parameters. Heart rate and respiration obtained from analogue outputs from standard clinical monitors or from specially designed hardware utilized routinely in the studies of human infants. The digitized recordings of ECG and respiration will be processed using software designed specifically for displaying, marking, and analyzing data from these records.
Change in Maternal Anxiety and Depressive Symptoms | Up to 12 months
  Mothers will complete various questionnaires measuring their mood and state.
Changes in Welch Emotional Connection Scale | Up to 12 months
  This is a clinical tool to assess the emotional connectedness of a mother-child dyad. The aim of the WECS is to assess behaviors observed during mother-child interaction, and score these behavioral observations across four domains to better inform health professionals of a dyad's interventional need. This scale will be completed by study staff.

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Welch, MD, Principal Investigator — Columbia University
Locations (1):
- Norwalk Housing Authority, Cos Cob, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Welch MG, Ludwig RJ, Hane AA, Austin J, Markowitz ES, Jaffe ME, Myers MM. Preschool-based mother-child emotional preparation program improves emotional connection, behavior regulation in the home and classroom: a randomized controlled trial. Front Child Adolesc Psychiatry. 2023 Oct 20;2:1232515. doi: 10.3389/frcha.2023.1232515. eCollection 2023. PMID 39816857